CLINICAL TRIAL: NCT03063866
Title: Randomised Controlled Study Comparing Use of Popofol Plus Fentanyl Versus Midazolam Plus Fentanyl as Sedation in Diagnostic Endoscopy in Patients With Advanced Liver Disease.
Brief Title: Randomised Controlled Study of Popofol Versus Midazolam as Sedation in Endoscopy With Advanced Liver Disease.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Consultant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Sameh 1
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- M group (Active Comparator): Midazolam 3 mg i.v added to fentanyl 0.5 ug/kg
  Interventions: Drug: Midazolam; Drug: Fentanyl
- P Group (Active Comparator): Propofol 1 mg/kg i.v added to fentanyl 0.5 ug/kg i.v
  Interventions: Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — Propofol 1 mg/kg i.v
  Other Names: propoven
  Arms: P Group
Drug: Midazolam — Midazolam 3 mg i.v
  Other Names: Dormicum
  Arms: M group
Drug: Fentanyl — fentanyl 0.5 ug/kg
  Other Names: Fantanyl

SUMMARY:
Gastrointestinal endoscopy is a frequent procedure in the patients with advanced liver disease. It requires variable degree of sedation ranging from minimal sedation to general anesthesia aiming for relieving pain, anxiety, and bad memories of the procedure.

In conscious sedation, patients are able to make purposeful responses to auditory and tactile clues, with maintenance of ventilatory and circulatory stability. while, in deep sedation, patients respond only to painful stimuli, and airway support is frequently required. At the level of general anesthesia, patients are unresponsive, and airway support is mandatory.

DETAILED DESCRIPTION:
The aim of this study is to compare use of propofol or midazolam as sedative for patients with advanced liver disease presented for gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40 and 60 years old.
* With Child score B or C
* Presented for elective gastrointestinal endoscopy

Exclusion Criteria:

* Emergent condition like hematemesis.
* Patients with moderate to severe hepatic encephalopathy.
* Patients with hepatopulmonary syndrome.
* Patients with known or suspected hypersensitivity to the used medication were also excluded from the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Level of sedation | 6 months
  Level of sedation using Ramsay sedation agitation score at before induction of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalek Ahmed, MD, Principal Investigator — Tanta University Faculty of Medicine; Sherief Abd-Elsalam, MD, Study Director — Tanta university Faculty of Medicine
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed SA, Selim A, Hawash N, Tawfik AK, Yousef M, Kobtan A, Badawi R, Elnawasany S, Elkhouly RA, Hanafy AS, Rizk FH, Mansour L, Abd-Elsalam S. Randomized Controlled Study Comparing Use of Propofol Plus Fentanyl versus Midazolam Plus Fentanyl as Sedation in Diagnostic Endoscopy in Patients with Advanced Liver Disease. Int J Hepatol. 2017;2017:8462756. doi: 10.1155/2017/8462756. Epub 2017 Sep 26. PMID 29312786